CLINICAL TRIAL: NCT04400227
Title: Pilot Study of Family Talk to Prevent Youth Substance Use
Brief Title: Preventing Youth Substance Use With Family Talk
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed due to change in funding.
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-38895; K23DA045085 (NIH)
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Substance Use Disorders
Keywords: parent-youth dyads; modules; prevention of adolescent SUD (substance use disorder); Family Talk
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Youth-Parent Dyads (Experimental): Participants will receive the Family Talk intervention and followup.
  Interventions: Other: Family Talk

INTERVENTIONS:
Other: Family Talk — Family Talk is an evidence-based, parent-youth dyadic approach that uses psychoeducation and skills building to help families make meaning of a parent's adversity, increase resilience, and improve family functioning.
  The Family Talk model comprises two components: the first involves a series of cognitive-behavioral techniques to bolster problem solving and communication skills among family members; the second involves a facilitated family meeting to develop a shared narrative for discussing each family member's experience of the parent's illness.

SUMMARY:
Family Talk, an evidence-based parent-youth dyadic intervention, is a promising approach to improving substance use outcomes for high-risk families, and its structure lends itself to delivery by existing personnel within an Office-Based Addiction Treatment (OBAT) model of care. The investigators propose a single-arm pilot study with 25 parent-youth dyads through which a rapid cycle performance improvement approach will be employed to adapt and optimize the content and delivery of the embedded Family Talk prevention strategy. The investigators will field-test relevant baseline and outcome measures and will use qualitative methodology to identify key modifications to the intervention and generate hypotheses for how the prevention strategy may impact youth and family outcomes and prevent youth substance use. Information from this study will inform a subsequent pilot randomized controlled trial of the intervention to prevent substance use for youth whose parents are in recovery from SUD (substance use disorder).

ELIGIBILITY:
Inclusion Criteria:

* Participating parent is receiving treatment for substance use disorder
* Participating youth is between the ages of 12-25
* Participating youth has no diagnosis of substance use disorder
* Parent and youth are both comfortable communicating in English or Spanish

Exclusion Criteria:

* Acute family crisis, such as recent or current incarceration, divorce, adult return to substance use, or traumatic event
* Adult or youth with cognitive limitation or intellectual disability

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in youth substance use based on the Timeline Followback Interview | baseline, 6 months
  The Timeline Followback Interview (TLFB) will be used to estimate substance use. It uses a calendar and asks the participant to indicate whether they used substances on each of the days listed for the last 3 months. No score is given for the measure. However, more days of use is associated with adverse health outcomes.
Youth substance use based on the Timeline Followback Interview at 2 months | 2 months
  The Timeline Followback Interview (TLFB) will be used to estimate substance use. It uses a calendar and asks the participant to indicate whether they used substances on each of the days listed for the last 3 months. No score is given for the measure. However, more days of use is associated with adverse health outcomes.
Youth substance use based on the Timeline Followback Interview at 4 months | 4 months
  The Timeline Followback Interview (TLFB) will be used to estimate substance use. It uses a calendar and asks the participant to indicate whether they used substances on each of the days listed for the last 3 months. No score is given for the measure. However, more days of use is associated with adverse health outcomes.
Change in Youth substance use based on the Screening to Brief Intervention Tool | baseline, 6 months
  The Screening to Brief Intervention instrument, or S2BI, is a 7-item instrument that asks about tobacco, alcohol, marijuana, prescribed drugs, inhalants, illegal drugs, and herbs/synthetic drugs. Responses for each substance can be 'never', 'once or twice', 'monthly', of 'weekly or more'. The result range from "no reported use," "lower risk," or "higher risk." For the lower and higher risk categories the intervention provides guidance for developing an action plan for each response category.
Youth substance use based on the Screening to Brief Intervention Tool at 2 months | 2 months
  The Screening to Brief Intervention instrument, or S2BI, is a 7-item instrument that asks about tobacco, alcohol, marijuana, prescribed drugs, inhalants, illegal drugs, and herbs/synthetic drugs. Responses for each substance can be 'never', 'once or twice', 'monthly', of 'weekly or more'. The result range from "no reported use," "lower risk," or "higher risk." For the lower and higher risk categories the intervention provides guidance for developing an action plan for each response category.
Youth substance use based on the Screening to Brief Intervention Tool at 4 months | 4 months
  The Screening to Brief Intervention instrument, or S2BI, is a 7-item instrument that asks about tobacco, alcohol, marijuana, prescribed drugs, inhalants, illegal drugs, and herbs/synthetic drugs. Responses for each substance can be 'never', 'once or twice', 'monthly', of 'weekly or more'. The result range from "no reported use," "lower risk," or "higher risk." For the lower and higher risk categories the intervention provides guidance for developing an action plan for each response category.

SECONDARY OUTCOMES:
Family Functioning based on the Family Problem Solving Communication Index | baseline, 2, 4, 6 months
  The Family Problem Solving Communication (FPSC) Index is a 10-item questionnaire designed to assess both positive and negative patterns of family communication. Answer choices are on a 4-point scale (0 = False, 1 = Mostly False, 2 = Mostly True and 3 = True). The two subscales can be scored separately, with Incendiary Communication measuring negative attributes and Affirmative Communication measuring positive forms of communication.
Family Functioning based on the Inventory of Parent and Peer Attachment | baseline, 2, 4, 6 months
  Inventory of Parent and Peer Attachment (IPPA) is a validated questionnaire that consists of 25 items for the mother, 25 items for the father, and 25 items for the adolescent. Three broad dimensions are assessed: degree of mutual trust, quality of communication, and extent of anger and alienation. Answers are rated on a 5-point Likert scale from 1 (almost never or never) to 5 (almost always or always). The IPPA is scored by reverse-scoring the negatively worded items and then summing the response values in each section.
Depression | baseline, 2, 4, 6 months
  Quick Inventory of Depressive Symptomatology is a 16-item questionnaire that measures rates of depression symptoms. Each answer in the survey is worth between 0 and 3 points. Severity of depression can be judged based on the total score. 1-5 = No depression 6-10 = Mild depression 11-15 = Moderate depression 16-20 = Severe depression 21-27 = Very severe depression.
Perceived Stress | baseline, 2, 4, 6 months
  Perceived Stress Scale (PSS) is a 10-item psychological instrument for measuring the perception of stress. Answer choices range from 0 to 4 (0=Never and 4=Very Often). PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items with higher scores indicating higher levels of stress.
Problem Solving | baseline, 2, 4, 6 months
  The Social Problem-Solving Inventory - Revised (SPSI-R) has both a long form (52 questions) and short form (25 questions) and assesses individual's strengths and weaknesses in their problem-solving abilities. The inventory has five component scales to assess problem-solving styles and solution generation: Positive Problem Orientation, Negative Problem Orientation, Rational Problem Solving, Impulsivity/Carelessness Style, Avoidance Style.
Coping based on the Coping Self-Efficacy Scale | baseline, 2, 4, 6 months
  The Coping Self-Efficacy Scale (CSES) is a 26-item measure of perceived self-efficacy for coping with challenges and threats. The answer choices are a rating on an 11-point scale. Anchor points on the scale are 0 ('cannot do at all'), 5 ('moderately certain can do') and 10 ('certain can do'). An overall CSES score is created by summing the item ratings with high scores indicate greater coping skills.
Coping based on the Brief COPE | baseline, 2, 4, 6 months
  The Brief COPE is a 28-item multidimensional measure of strategies used for coping or regulating cognitions in response to stressors. There are 14 two-item subscales within the Brief COPE, and each is analyzed separately: (1) self-distraction, (2) active coping, (3) denial, (4) substance use, (5) use of emotional support, (6) use of instrumental support, (7) behavioral disengagement, (8) venting, (9) positive reframing, (10) planning, (11) humor, (12) acceptance, (13) religion, and (14) self-blame. Respondents rate items on a 4-point Likert scale, ranging from 1 - "I haven't been doing this at all" to 4 - "I've been doing this a lot." Each of the 14 scales is comprised of 2 items; total scores on each scale range from 2 (minimum) to 8 (maximum). Higher scores indicate increased utilization of that specific coping strategy.
Social support | baseline, 2, 4, 6 months
  The Social Adjustment Scale-Self-Report (SAS-SR) 54-item measure that evaluates the efficacy of pharmacological treatments of mental disorders to provide an understanding of a client's satisfaction with his or her social situation. Answer choices are on a 5-point Likert scale with higher scores indicating a better quality of life.
Stressful Life Events | baseline, 2, 4, 6 months
  The Stressful Life Events Screening Questionnaire (SLESQ) is a 13-item self-report measure that assesses lifetime exposure to traumatic events. For each event, respondents are asked to indicate whether the event occurred ("yes" or "no"), their age at time of the event, as well as other specific items related to the event, such as the frequency, duration, whether anyone died, or was hospitalization, etc. No score is given for the measure.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Kistin, MD MSc, Principal Investigator — Boston Medical Center; Scott Hadland, MD, Study Director — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No